CLINICAL TRIAL: NCT04030338
Title: Serial PSMA PET Imaging in the Assessment of Treatment Response in Patients With Progressive Prostate Cancer
Brief Title: Prostate-Specific Membrane Antigen (PSMA) PET Scans in People Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-170
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Prostate Neoplasm; Prostate Adenocarcinoma; Prostate Cancer Metastatic; Metastatic Prostate Cancer
Keywords: prostate cancer; Metastatic Prostate Cancer; PCWG3; 18 F-DCFPyL; 68 Ga-PSMA; 19-170; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate cancer: Participants with histologically confirmed prostate cancer, that is either newly diagnosed OR progressive as defined by standard PCWG3 criteria. Patients w ill remain on study until 30 days after their last PSMA imaging timepoint required by their companion therapeutic protocol.
  Interventions: Drug: 18F-DCFPyL-iPSMA; Drug: 68Ga-HBED-iPSMA; Diagnostic Test: PET/CT scan

INTERVENTIONS:
Drug: 18F-DCFPyL-iPSMA — Participants will be injected intravenously with a bolus of 7-10 mCi of 18F-DCFPyL.
Drug: 68Ga-HBED-iPSMA — Participants will be injected intravenously with a bolus of 3-8 mCi of 68Ga-HBED-iPSMA
Diagnostic Test: PET/CT scan — The baseline PSMA PET scan may be performed externally or at MSKCC, but all follow-up imaging must be performed at MSKCC. Approximately 60-90 minutes after intravenous injection of radiotracer, patients will be scanned from the mid-skull to the mid-thigh. Imaging will start with a low-dose CT for attenuation correction, followed by a PET scan. Upon completion of imaging and at the discretion of the investigator, the patient may be asked to void and get back in the scanner for 1 additional image of the pelvis.This additional image allows investigator's to see an unobstructed view of the prostate/prostate bed

SUMMARY:
The purpose of this study is to determine if Prostate-Specific Membrane Antigen (PSMA) positron emission tomography (PET) scans used in this study accurate and better at imaging participants' prostate cancer than the usual methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed prostate cancer, that is either: newly diagnosed OR progressive as defined by standard PCWG3 criteria. note that metastatic disease is defined by either bone scintigraphy or by CT or MRI, or a combination of these tests, but not exclusively by molecular imaging criteria.

Patients with newly diagnosed localized or metastatic prostate cancer are eligible, provided standard imaging (either bone scintigraphy, CT or MRI) demonstrates evidence of radiographic disease

Patient with progressive disease that is non-metastatic are eligible by biochemical progression: A minimum of three rising PSA values from a baseline that are obtained 1 week or more apart, or 2 measurements 2 or more weeks apart

Patients with progressive disease that is metastatic are eligible either by biochemical progression or radiographic progression or both

Patients are permitted to have had up to 2 months of prior hormonal therapy before entering this trial (and many therapeutic trials) and therefore, their progression criteria would apply to their pre-treatment imaging and PSA parameters Note: This criterion pertains to patients with newly diagnosed, untreated disease. This criterion does not apply to those who were already on therapy for metastatic CRPC.

* Karnofsky performance status of >/= 50 (or ECOG/WHO equivalent)
* Male (or transgender female) > 18 years of age
* Patient must be able to understand and willing to sign a written informed consent document
* Patient is anticipating starting a therapeutic strategy following imaging

Exclusion Criteria:

* Patient undergoing active treatment for non-prostate malignancy, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and non-invasive bladder cancer
* Unable to lie flat, still or tolerate a PET scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan Kettering Cancer Center (MSK) in the Department of Medical Oncology, Radiology, Radiation Oncology or Surgery. Investigators will screen their patients' medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Measure predictive accuracy of the change in PSMA PET with respect to the time to biochemical progression | start of treatment to the first PSA level above 0.2 ng/ml, up to 100 months
Measure predictive accuracy of the change in PSMA PET with respect to the time to metastasis | Time from the start of treatment to evidence of systemic disease on bone scan or CT/MRI, up to 100 months
Measure predictive accuracy of the change in PSMA PET with respect to overall survival time. | Time from the start of treatment to date of death from any cause, assessed up to up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schoder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT04030338/ICF_000.pdf